CLINICAL TRIAL: NCT01579240
Title: Internet Intervention Promotes Physical Activity
Brief Title: Internet Intervention Promotes Physical Activity in Sedentary Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, A. Blair Irvine, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SBIR51 Sr. Exercise; R44AG020002 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2006-12

CONDITIONS: Exercise; Sedentary Older Adults
Keywords: physical activity; older adults; Internet; sedentary; multi-week; internet intervention
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- program visits (Experimental): visits to intervention program
  Interventions: Other: Internet exercise program

INTERVENTIONS:
Other: Internet exercise program — 12 voluntary weekly visits to website

SUMMARY:
This study evaluated the efficacy of a 12-week Internet intervention to help sedentary older adults adopt and maintain an exercise regimen. A total of 368 men and women over 55 years of age (x = 60.3; SD 4.9 ) were recruited and screened on line. They randomized into treatment and control groups and assessed at pre-test, 12 weeks, and at six months.

The multivariate model was significant at posttest (p = .001; large effect size) and at six months (p = .001; medium effect size). At posttest, intervention participation showed significant improvement on 13 of 14 outcome measures compared to the control group. At six months, treatment group participants were found to maintain large gains compared to the Ctrl participants on all 14 measures.

DETAILED DESCRIPTION:
Based on the treatment group users self reported fitness level, activity goals, and self-identified barriers to exercise, the program helped users select exercise activities in the areas of endurance, flexibility, strengthening, and balance enhancement. They returned weekly for automated video and text support and education, with the option to change or increase in their exercise plan, and on-going problem solving to overcome barriers to exercise.

ELIGIBILITY:
Inclusion Criteria:

* > 54 years of age;
* < 61 minutes of exercise per week;
* internet connection; email address

Exclusion Criteria:

* too young;
* too active;
* no web access;
* no email

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2006-02; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular exercise | Baseline-6 months
  Self report: minutes/week

SECONDARY OUTCOMES:
Psycho-social measures (attitudes, knowledge, self efficacy, intentions) | Baseline - 6 months.
  Self rated survey items

CONTACTS AND LOCATIONS:
Locations (1):
- ORCAS, Eugene, Oregon, United States